CLINICAL TRIAL: NCT07324980
Title: Acute Dyspnea in the Emergency Department: Diagnostic Evaluation of Inferior Vena Cava Ultrasound Integrated With Multimodal Point-of-Care Ultrasound and Clinical Data
Brief Title: Acute DYSPnea in the Emergency Department: Diagnostic Value of Point-of-care UltraSound
Acronym: DYSP-ED-US
Status: Recruiting | Type: Observational
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Francesco Gavelli, Emergency Medicine Associate Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: CE218/2025
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hydrostatic Pulmonary Edema; Acute Respiratory Failure; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute dyspnea is a common reason for emergency department (ED) admission and is frequently caused by acute heart failure with pulmonary edema. Rapid differentiation between cardiogenic and non-cardiogenic causes of dyspnea is essential to guide early treatment and risk stratification. However, no single gold standard exists for the assessment of venous congestion in the acute setting.

This prospective observational study aims to evaluate the diagnostic accuracy of respiratory variation in inferior vena cava (IVC) diameter measured by point-of-care ultrasound (POCUS) in identifying acute pulmonary edema in patients presenting to the ED with acute respiratory failure. In addition, the study investigates whether integration of IVC ultrasound with lung ultrasound, bedside cardiac ultrasound, and selected clinical and laboratory variables - such as hemoglobin and plasma protein changes - improves diagnostic performance and prognostic stratification.

DETAILED DESCRIPTION:
Acute heart failure is a leading cause of emergency department visits and hospital admissions and is associated with high morbidity, mortality, and healthcare costs. Dyspnea is the most frequent presenting symptom. Early identification of pulmonary edema and assessment of venous congestion are critical to optimize therapeutic decisions in the acute phase.

Ultrasound assessment of inferior vena cava (IVC) respiratory variation has been proposed as a rapid, non-invasive marker of volume overload and venous congestion. However, its reliability during the early stages of acute dyspnea remains uncertain, particularly in patients with increased respiratory effort. Other ultrasound-based approaches, including lung ultrasound, and focused cardiac ultrasound, provide complementary information on pulmonary congestion and cardiac function.

This single-center, prospective, observational study will enroll adult patients presenting to the emergency department with acute dyspnea and respiratory failure. All participants will undergo standardized clinical assessment, laboratory testing, chest imaging as per routine care, and multimodal point-of-care ultrasound evaluation at ED admission, after 1 hour, and at 24-48 hours when clinically feasible.

The primary objective is to assess the diagnostic accuracy of respiratory variation in IVC diameter for identifying acute pulmonary edema. Secondary objectives include evaluation of multimodal ultrasound-clinical scores for diagnostic and prognostic purposes and analysis of early changes in hemoglobin and plasma proteins as surrogate markers of fluid shifts. Clinical outcomes, including need for hospitalization, escalation of care, and in-hospital mortality, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Presentation to the emergency department with acute dyspnea and acute respiratory failure, defined by at least one of the following:

  * PaO₂ < 60 mmHg on room air, or
  * Oxygen saturation (SpO₂) < 90% on room air, or
  * PaO₂/FiO₂ ratio < 300.
* Ability to provide written informed consent or eligibility for deferred consent according to local regulations.
* Undergoing standard diagnostic evaluation including laboratory tests and chest imaging as part of routine clinical care.

Exclusion Criteria:

* Refusal to provide informed consent (or consent by legal representative when applicable).
* Inadequate ultrasound window or technically insufficient ultrasound assessment.
* Acute respiratory failure secondary to chest trauma.
* Cardiac arrest at presentation or during emergency department stabilization.
* Requirement for invasive mechanical ventilation during initial stabilization in the emergency department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the emergency department with acute dyspnea and acute respiratory failure, undergoing standard diagnostic evaluation and clinical management as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of respiratory variation in inferior vena cava (IVC) diameter for acute pulmonary edema | At emergency department admission (baseline, T0) and after 1 hour (T1)
  Diagnostic performance of respiratory variation in inferior vena cava diameter, measured by point-of-care ultrasound (POCUS), in discriminating acute pulmonary edema from other causes of acute dyspnea in the emergency department.

SECONDARY OUTCOMES:
Diagnostic performance of early changes in hemoglobin concentration | At emergency department admission (baseline, T0) and after 1 hour (T1)
  Diagnostic performance of early variation in hemoglobin concentration - as a surrogate marker of fluid shifts - in discriminating acute pulmonary edema from other causes of acute dyspnea in the emergency department
Diagnostic performance of early changes in plasma protein concentration | At emergency department admission (baseline, T0) and after 1 hour (T1)
  Diagnostic performance of early variation in plasma protein concentration - as a surrogate marker of fluid shifts - in discriminating acute pulmonary edema from other causes of acute dyspnea in the emergency department.

OTHER OUTCOMES:
Diagnostic performance of multimodal ultrasound-clinical integration | At emergency department admission (baseline, T0) and after 1 hour (T1)
  Diagnostic accuracy of integrated multimodal assessment combining inferior vena cava ultrasound, lung ultrasound, focused cardiac ultrasound, and selected clinical and laboratory variables for the diagnosis of acute pulmonary edema.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No
Results are reported only in aggregated form.

REFERENCES:
- [Background] Gavelli F, Castello LM, Monnet X, Azzolina D, Nerici I, Priora S, Via VG, Bertoli M, Foieni C, Beltrame M, Bellan M, Sainaghi PP, De Vita N, Patrucco F, Teboul JL, Avanzi GC. Decrease of haemoconcentration reliably detects hydrostatic pulmonary oedema in dyspnoeic patients in the emergency department - a machine learning approach. Int J Emerg Med. 2024 Sep 5;17(1):114. doi: 10.1186/s12245-024-00698-y. PMID 39237860